CLINICAL TRIAL: NCT03735355
Title: Endoscopic Balloon Dilation as Compared to Surgical Management for the Treatment of Short Strictures in Fibrostenosing Crohns Disease: A Randomized Controlled Trial.
Brief Title: Endoscopic Balloon Dilation vs Surgery to Treat Short Strictures in Fibrostenosing Crohns Disease: An RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Mohammad Yaghoobi, Assistant Professor of Medicine, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TTS Surgery Crohns Stricture
Record Dates: First submitted 2018-11-05; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balloon dilation (Experimental): TTS balloon dilation
  Interventions: Procedure: TTS balloon dilation
- Surgery (Active Comparator): Resection of the fibrostenotic area
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — Surgical resection of fibrostenotic area
  Arms: Surgery
Procedure: TTS balloon dilation — Dilation of a stricture using TTS balloon
  Arms: Balloon dilation

SUMMARY:
There is currently no standard management to guide the clinicians in treating patients with fibrostenotic disease. European Crohns and Colitis Organization [ECCO] recently developed a topical review on prediction, diagnosis and management of fibrostenosing Crohns disease. The review suggests endoscopic balloon dilation, strictureplasty, and intestinal resection as reasonable treatment options for short strictures based on the low grade of evidence.

DETAILED DESCRIPTION:
Study Population All patients with Crohns disease and a short stricture (<5 cm) within the reach of upper or lower GI endoscopy

Study Timeline

1. Pre-recruitment phase including proposal, IRB approval, staff training, budget transfer - 9 months
2. Recruitment of patients: 2 years
3. Follow up: 2 years
4. Analysis and preparing report: 6 months

Study Design Single blind randomized controlled trial The data will be blindly analyzed. Double blinding is not possible due to the nature of the study.

Study Methods Please see the study flow diagram below. Randomization will be done using computer software generating random numbers. Outcome Measures - A research associate will contact patients on weeks 1,2,4 and months 3,6,12,18 and 24 to record the items mentioned as secondary objectives of the study.

- An interim analysis will be performed after 20 cases complete the study Sample Size 40 patients randomized to two arms undergoing TTS dilation or surgical managements

Statistical analysis Comparisons between groups will be done using Student's t-test. Qualitative variables will be summarized as a percentage of the group total and comparisons between groups will be based on the chisquared test. The cumulative relapse rate of each treatment group will be estimated by the Kaplan±Meier method and the difference between treatment groups will be tested by the log rank test. Time to relapse will be compared betweens two groups using a Cox proportional hazards regression analysis. A P value of less than 0.05 is considered to be signicant.

ELIGIBILITY:
Inclusion Criteria:

* 40 Patients with Crohns disease and a short stricture (<5 cm) within the reach of upper or lower GI endoscopy

Exclusion Criteria:

* Abscess or phlegmon
* Fistula
* High-grade dysplasia
* Malignancy
* Previous intervention
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Surgery-free period in patients with fibrostenotic Crohns disease | 2 years
  The time to the need for first surgical treatment in following study intervention in each group

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rieder F, Latella G, Magro F, Yuksel ES, Higgins PD, Di Sabatino A, de Bruyn JR, Rimola J, Brito J, Bettenworth D, van Assche G, Bemelman W, d'Hoore A, Pellino G, Dignass AU. European Crohn's and Colitis Organisation Topical Review on Prediction, Diagnosis and Management of Fibrostenosing Crohn's Disease. J Crohns Colitis. 2016 Aug;10(8):873-85. doi: 10.1093/ecco-jcc/jjw055. Epub 2016 Feb 29. PMID 26928961